CLINICAL TRIAL: NCT03669913
Title: Mitigating Adverse Sexual and Reproductive Health Outcomes Through a Comprehensive Primary School Sexuality Education Program in South-Western Uganda
Brief Title: Mitigating Adverse Sexual and Reproductive Health Outcomes Among Young Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: University Ghent (Other); Free University of Brussels (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MUST 04/10-15
Record Dates: First submitted 2018-09-07; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Relationship Problems Specific to Childhood and Adolescence
Keywords: sexuality; education; adolescents
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Intervention Model Description: A cluster randomized trial where the intervention is structured comprehensive sexuality education lesson packages
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention arm will receive a pre evaluation survey, 11 lessons on CSE sequentially in a period of one year and a post evaluation survey
  Interventions: Other: Lessons on comprehensive sexuality education
- Control arm (No Intervention): This is a control arm that receives no intervention but will have and pre and post evaluation in one year

INTERVENTIONS:
Other: Lessons on comprehensive sexuality education — Provision of 11 standardized lessons on comprehensive sexuality education based on international guidance on sexuality education by UNESCO
  Arms: Intervention

SUMMARY:
This study evaluates the effectiveness of comprehensive sexuality education (CSE) among young adolescents (10-14 years) in schools. A total of 33 schools will participate in the trial with 15 intervention arm that will receive CSE education and 18 in the control arm, Intervention will go on for one year

DETAILED DESCRIPTION:
The International Technical Guidance on Sexuality Education (ITGSE) defines CSE as "an age-appropriate, culturally relevant approach to teaching about sexuality and relationships by providing scientifically accurate, realistic, non-judgmental information and CSE improves sexual and reproductive health outcomes of young people by delaying sexual debut, promoting condom use and increasing sexual health knowledge, however, most of these outcomes have been reported in older adolescents and there is limited evidence for effectiveness of CSE among young adolescents

The study aims at improving adolescent sexual and reproductive health of young adolescents through CSE that is led by interdisciplinary university students' team in an environment where no consistent or regulated sexual and reproductive health education program currently exists

ELIGIBILITY:
Inclusion Criteria:

* adolescent 10-14 years in primary school
* Adolescent in primary 5 or 6 of education in Uganda
* Written consent/assent to participate

Exclusion Criteria:

* Below 10 years or above 14 years at baseline
* No consent obtained

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1100 (Estimated)
Dates: Start 2015-11-08 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
change in sexual health knowledge by 15% from baseline | one year
  change in sexual health knowledge(HIV, STI, contraception and puberty knowledge) using an itemized questionnaire developed for the study. The estimated knowlege score will be 25 . Individual items include on knowledge of puberty, HIV/STIs and pregnancy prevention. This includes knowledge on how HIV/AIDS can be acquired (score 0-4), types of common Sexually Transmitted Infections (score 0-4), knowledge of pubertal changes in boys (score 0-6.) and in girls (score 0-7), and knowledge about ways to prevent pregnancy (score 0-4)

SECONDARY OUTCOMES:
Change in proportion of sexually active adolescents by 10% from baseline | one year
  Change in number of those who are sexually active
Change in gender equitable norm scores by 10% from baseline | one year
  Adolescents to adopt a more gender equitable norm attitude. Gender equitable norms scale will be developed on a 4 likert point scale and total scores will range from 0 to 44. The higher the score, the higher the tendency to have gender equitable norms. The score consists of 11 items. Six of these items were adapted from the Attitudes towards Women Scale for Adolescents (AWSA) by Galambos NL et al., 1985 while 5 items were developed to suit the respondents' age and the Ugandan context.
change in body image scores by 10% from baseline | one year
  Adolescents develop a more positive attitude in appreciation of their body size or shape.The items for this scale were adapted from the Body Image States Scale (BISS-6) by Cash TF et al, 2002 but transformed to a 5 point likert scale including a neutral point for ease of use among respondents. The total expected score was 24 and the higher the score the better the body image
change in self esteem scores by 10% from baseline | one year
  Adolescent develop confidence in themselves and their abilities. Self esteem score used was developed by Rosenberg M et al., 1965. The total expected score for the 10 items was 40. The higher the score the better the self esteem

CONTACTS AND LOCATIONS:
Overall Officials: Kristien Michielsen, PhD, Principal Investigator — University Ghent

IPD SHARING:
Plan to Share IPD: Undecided
Data will be discretely shared with other researchers on request

REFERENCES:
- [Background] Rosenberg M. Rosenberg self-esteem scale (RSE). Acceptance and commitment therapy. Measures package. 1965;61:52.
- [Background] Cash TF, Fleming EC, Alindogan J, Steadman L, Whitehead A. Beyond body image as a trait: the development and validation of the Body Image States Scale. Eat Disord. 2002 Summer;10(2):103-13. doi: 10.1080/10640260290081678. PMID 16864251
- [Background] Galambos NL, Petersen AC, Richards M, Gitelson IB. The Attitudes Toward Women Scale for Adolescents (AWSA): A study of reliability and validity. Sex roles. 1985;13(5):343-356.
- [Background] Kemigisha E, Nyakato VN, Bruce K, Ndaruhutse Ruzaaza G, Mlahagwa W, Ninsiima AB, Coene G, Leye E, Michielsen K. Adolescents' Sexual Wellbeing in Southwestern Uganda: A Cross-Sectional Assessment of Body Image, Self-Esteem and Gender Equitable Norms. Int J Environ Res Public Health. 2018 Feb 22;15(2):372. doi: 10.3390/ijerph15020372. PMID 29470388

DOCUMENTS (1):
  • Study Protocol (2016-11-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT03669913/Prot_000.pdf